CLINICAL TRIAL: NCT04394624
Title: Open-label, Single-arm Trial to Evaluate Antitumor Activity, Safety, and Pharmacokinetics of Tusamitamab Ravtansine (SAR408701) Used in Combination With Ramucirumab or Ramucirumab and Pembrolizumab in Metastatic, Non-squamous, Non Small-cell Lung Cancer (NSQ NSCLC) Patients With CEACAM5-positive Tumors, Previously Treated With Platinum-based Chemotherapy and an Immune Checkpoint Inhibitor
Brief Title: Tusamitamab Ravtansine (SAR408701) in Combination With Ramucirumab or Ramucirumab and Pembrolizumab in Pretreated Patients With NSQ NSCLC (CARMEN-LC04)
Acronym: CARMEN-LC04
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision, the decision is not related to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT16525; U1111-1244-1585 (Registry Identifier: ICTRP); 2019-003914-15 (EudraCT Number)
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer Metastatic
MeSH Terms: interventions — tusamitamab ravtansine; Ramucirumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ramucirumab + SAR408701 (Experimental): Ramucirumab will be administered intravenously prior to intravenously adminstration of SAR408701 every two 2 weeks.
  Interventions: Drug: SAR408701; Drug: ramucirumab
- Ramucirumab + pembrolizumab +SAR408701 (Experimental): Participants will be treated with tusamitamab ravtansine and ramucirumab and pembrolizumab to assess the tolerability of the combination
  Interventions: Drug: SAR408701; Drug: ramucirumab; Drug: pembrolizumab

INTERVENTIONS:
Drug: SAR408701 — Pharmaceutical form:concentrate for solution for injection Route of administration: intravenous infusion
Drug: ramucirumab — Pharmaceutical form: concentrate for solution for injection Route of administration: intravenous infusion
Drug: pembrolizumab — Pharmaceutical form: concentrate for solution for injection Route of administration: intravenous infusion
  Arms: Ramucirumab + pembrolizumab +SAR408701

SUMMARY:
Primary Objectives:

Doublet Cohort

Part 1 (safety run-in):

To assess the tolerability and to confirm the recommended dose of tusamitamab ravtansine in combination with ramucirumab in the NSQ NSCLC population.

Part 2:

To assess the antitumor activity of tusamitamab ravtansine in combination with ramucirumab in the NSQ NSCLC population.

Triplet cohort

To assess the tolerability and to confirm the recommended dose of tusamitamab ravtansine in combination with ramucirumab and pembrolizumab in the NSQ NSCLC population.

Secondary Objectives:

Doublet Cohort

To assess the safety and tolerability of tusamitamab ravtansine in combination with ramucirumab.

To assess the durability of the response to treatment with tusamitamab ravtansine in combination with ramucirumab.

To assess anti-tumor activity of tusamitamab ravtansine in combination with ramucirumab on progression free survival (PFS) and disease control rate (DCR).

To assess the pharmacokinetic (PK) profiles of tusamitamab ravtansine (SAR408701) and ramucirumab when given in combination.

To assess the immunogenicity of tusamitamab ravtansine (SAR408701) when given in combination with ramucirumab.

Triplet cohort

To assess the safety and tolerability of tusamitamab ravtansine in combination with ramucirumab and pembrolizumab

To assess the antitumor activity of tusamitamab ravtansine in combination with ramucirumab and pembrolizumab in the NSQ NSCLC population.

To assess the immunogenicity of tusamitamab ravtansine when given in combination with ramucirumab and pembrolizumab

DETAILED DESCRIPTION:
The expected duration of the study intervention for participants may vary, based on progression date ; median expected duration of study per participant is estimated 11 months (up to 1 month for screening, a median of 6 months for treatment, and a median of 4 months for end-of-treatment assessments and safety follow-up visit)

ELIGIBILITY:
Inclusion criteria :

* Metastatic disease progression fulfilling both of the following 2 criteria:

  1. Having progressive disease during or after platinum-based chemotherapy (at least 2 cycles). Maintenance therapy following platinum-based chemotherapy is not considered as a separate regimen. Adjuvant/neoadjuvant treatment for a patient who had a relapse with metastatic disease during or within 6 months of completing treatment will be considered as first-line treatment.

     AND
  2. Having progressive disease during or after 1 immune checkpoint inhibitor (anti-PD1/PD-L1); this could be given as monotherapy or in combination with platinum-based chemotherapy (whatever the order).
* Participants with carcinoembryonic antigen-related cell adhesion molecule (CEACAM) 5 expression of ≥2+ in archival tumor sample (or if not available, fresh biopsy sample) involving at least 50 % of the tumor cell population as demonstrated prospectively by central laboratory via immune histochemistry (IHC).
* At least one measurable lesion by RECIST v1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* A female participant who agrees to use effective contraceptive methods during and for at least 7 months after the last dose of study intervention.
* A male participant who agrees to use effective contraception methods during and for at least 4 months after the last dose of study intervention
* Signed informed consent

Exclusion criteria:

Participants are excluded from the study if any of the following criteria apply:

* Patients with untreated brain metastases and history of leptomeningeal disease.
* Significant concomitant illnesses that would impair the patient's participation in the study or interpretation of the results.
* History within the last 3 years of an invasive malignancy other than the one treated in this study, with the exception of resected/ablated basal or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix, or other local tumors considered cured by local treatment.
* Non-resolution of any prior treatment related toxicity to < grade 2 according to NCI CTCAE V5.0, except for alopecia, vitiligo and active thyroiditis controlled with hormonal replacement therapy
* History of known acquired immunodeficiency syndrome (AIDS) related illnesses or known HIV disease requiring antiretroviral treatment, or unresolved viral hepatitis
* Previous history of and/or unresolved corneal disorders. The use of contact lenses is not permitted.
* Radiographic evidence of major airway or blood vessel invasion or intratumor cavitation
* History of uncontrolled hereditary or acquired arterial thrombotic disorder or history of aneurism.
* Major surgery within 28 days prior to Day 1/first IMP infusion,. Postoperative bleeding complications or wound complications from a surgical procedure performed in the last 2 months.
* History of gross hemoptysis within 2 months before the first administration of study intervention.
* Clinically relevant congestive heart failure (CHF; NYHA II-IV, or LVEF less than 50%) or symptomatic or poorly controlled cardiac arrhythmia.
* Any arterial thrombotic event within 6 months before the first administration of study intervention.
* Uncontrolled arterial hypertension (systolic ≥150 mmHg or diastolic ≥90 mmHg) despite standard medical management.
* Serious or nonhealing wound, skin ulcer, or bone fracture within 28 days before the first administration of study intervention.
* Gastrointestinal (GI) perforation and/or fistulae within 6 months prior to first administration of study intervention.
* Significant bleeding disorders, vasculitis, or Grade 3-4 gastrointestinal (GI) bleeding within 3 months before the first administration of study intervention.
* Bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection Crohn's disease, ulcerative colitis, or chronic diarrhea.
* Medical condition requiring concomitant administration of a medication with a narrow therapeutic window and metabolized by CYP450 or a strong CYP3A inhibitor
* Concurrent treatment with any other anticancer therapy
* No more than 1-line previous chemotherapy in metastatic setting
* Prior treatment with ramucirumab or docetaxel
* Prior therapy targeting CEACAM5 or maytansinoid treatment (DM1 or DM4 antibody-drug conjugate)
* Contraindication to use of corticosteroid premedication
* Current therapeutic anticoagulation with warfarin, low-molecular-weight heparin, or similar agents. Patients receiving prophylactic, low-dose anticoagulation therapy are eligible
* Previous enrollment in this study, current participation in any other clinical study involving an investigational study treatment, or any other type of medical research
* Poor bone marrow, liver or kidney functions
* Urine dipstick or routine analysis indicating proteinuria of 2+ or higher, unless a 24 hour urine collection demonstrates <1000 mg of protein.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.Most important exclusion criteria for potential participants

Triplet cohort exclusions

* History of active autoimmune disease that has required systemic treatment in the past 2 years.
* History of allogeneic tissue/solid organ transplantation.
* Active infection requiring IV systemic therapy within 2 weeks prior to first study intervention administration or active tuberculosis.
* Interstitial lung disease or history of pneumonitis that has required oral or IV steroids.
* Symptomatic herpes zoster within 3 months prior to screening.
* Significant allergies to humanized monoclonal antibodies.
* Any radiation therapy to lung >30 Gy within 6 months of first study intervention administration.
* Has received or will receive a live vaccine within 30 days prior to the first study intervention administration.
* Thyroid-stimulating hormone (TSH) out of normal limits. If TSH is not within normal limits at baseline, the subject may still be eligible if T3 and free T4 are within the normal limits

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2024-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- United States (3):
  - Henry Ford Hospital Site Number : 8400005, Detroit, Michigan
  - Roswell Park Cancer Institute Site Number : 8400003, Buffalo, New York
  - McClinton Cancer Center Site Number : 8400002, Waco, Texas
- Investigational Site Number : 1000001, Plovdiv, Bulgaria
- Czechia (2):
  - Investigational Site Number : 2030001, Ostrava - Vitkovice
  - Investigational Site Number : 2030002, Prague
- Investigational Site Number : 6200001, Porto, Portugal
- South Korea (2):
  - Investigational Site Number : 4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (4):
  - Investigational Site Number : 7240001, Barcelona / Sabadell, Catalunya [Cataluña]
  - Investigational Site Number : 7240005, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240004, Madrid
  - Investigational Site Number : 7240003, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 centers in 5 countries. A total of 37 participants were screened between 31 August 2020 and 03 October 2022, of which 6 were screen failures. Screen failures were mainly due to not meeting the criteria for inclusion. The study was prematurely terminated due to the discontinuation of the overall development of tusamitamab ravtansine (SAR408701) by the sponsor.
Pre-assignment Details: A total of 31 participants were enrolled in the study. No participants were enrolled in the triplet cohort due to the early termination of the study.
Groups:
- Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab: Participants received tusamitamab ravtansine 100 milligram per square meter (mg/m^2) and ramucirumab 8 mg per kilogram (kg) intravenous (IV) infusion every 2 weeks (Q2W) until disease progression, unacceptable adverse event (AE), or the participant's or investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab: Participants were planned to receive tusamitamab ravtansine 150 mg/m^2 plus ramucirumab 10 mg/kg and pembrolizumab 200 mg IV infusion every 3 weeks (Q3W) until disease progression, unacceptable AE, or the participant's or investigator's decision to stop the treatment.
Period: Overall Study
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Started | 31 | 0
Completed (Treatment completed) | 0 | 0
Not Completed | 31 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Progressive disease | 24 | 0
Not completed — Not related to COVID-19 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered. No participants were enrolled in the triplet cohort due to the early termination of the study.
Groups:
- Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab: Participants received tusamitamab ravtansine 100 mg/m^2 and ramucirumab 8 mg/kg IV infusion Q2W until disease progression, unacceptable AE, or the participant's or investigator's decision to stop the treatment.
- Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab: Participants were planned to receive tusamitamab ravtansine 150 mg/m^2 plus ramucirumab 10 mg/kg and pembrolizumab 200 mg IV infusion Q3W until disease progression, unacceptable AE, or the participant's or investigator's decision to stop the treatment.
- Total: Total of all reporting groups
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab | Total
Number analyzed (Participants) | 31 | 0 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (10.1) |  | 62.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 |  | 16
  Male | 15 |  | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 13 |  | 13
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 18 |  | 18
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study drug, whether or not considered related to the study drug. A SAE is defined as any untoward medical occurrence that, at any dose: results in death or life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization or results in persistent disability/incapacity or congenital anomaly/birth defect. TEAE is defined as AEs that develop, worsen, or become serious during the treatment period.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants
  Any TEAE | 31 |
  Any treatment-emergent SAE | 7 |

2. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Hematology
Description: Blood samples were collected to determine the hematology laboratory clinically significant abnormalities.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered. Only those participants with data collected are reported. No participants were enrolled in the triplet cohort due to the early termination of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants
  Anemia | 19 |
  White blood cell decreased | 8 |
  Neutrophil count decreased | 8 |
  Lymphocyte count decreased | 11 |
  Eosinophilia | 12 |
  Platelet count decreased | 21 |
  International normalized ratio increased | 2 |
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 30 | 0
  Activated partial thromboplastin time prolonged | 11 |

3. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Metabolism
Description: Blood samples were collected to determine the clinically significant abnormalities in metabolism.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants
  Hypoglycemia | 1 |
  Hypoalbuminemia | 16 |
  Total protein: <Lower limit of normal | 3 |
  Total protein: >Upper limit of normal | 4 |

4. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Electrolytes
Description: Blood samples were collected to determine the clinically significant abnormalities in electrolytes.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants
  Hyponatremia | 15 |
  Hypernatremia | 2 |
  Hypokalemia | 7 |
  Hyperkalemia | 9 |
  Hypocalcemia | 6 |
  Hypercalcemia | 5 |

5. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Renal Function
Description: Blood samples were collected to determine the renal function laboratory clinically significant abnormalities.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants | 10 |

6. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Liver Function
Description: Blood samples were collected to determine the liver function laboratory clinically significant abnormalities.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants
  Alanine aminotransferase increased | 19 |
  Aspartate aminotransferase increased | 21 |
  Alkaline phosphatase increased | 12 |
  Blood lactate dehydrogenase increased | 26 |
  Total bilirubin increased | 6 |

7. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Electrocardiogram (ECG)
Description: A single 12-lead ECG was recorded using an ECG machine that automatically calculates the heart rate and measures PR, QRS, and QT intervals.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants
  Heart Rate: >90 beats per minute (bpm) | 22 |
  Heart Rate: >90 bpm and increase from baseline >=20 bpm | 13 |
  Heart Rate: >100 bpm | 14 |
  Heart Rate: >100 bpm and increase from baseline >=20 bpm | 8 |
  Heart Rate: >120 bpm | 1 |
  PR Interval: >200 milliseconds (msec) | 4 |
  PR Interval: >200 msec and increase from baseline >=25% | 1 |
  PR Interval: >220 msec | 2 |
  PR Interval: >220 msec and increase from baseline >=25% | 1 |
  QRS Interval: >110 msec | 6 |
  QRS Interval: >110 msec and increase from baseline >=25% | 1 |
  QRS Interval: >120 msec | 2 |
  QT Interval: >500 msec | 1 |
  QTcF Prolongation: >450 msec | 8 |
  QTcF Prolongation: >480 msec | 2 |
  QTcF Prolongation: >500 msec | 1 |
  QTcF Prolongation: Increase from baseline [30-60] msec | 9 |
  QTcF Prolongation: Increase from baseline >60 msec | 2 |

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities: Urinalysis
Description: Urine samples were collected to determine the clinically significant abnormalities in urine.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants
  Urine Protein: Negative | 8 |
  Urine Protein: + | 12 |
  Urine Protein: ++ | 3 |
  Urine Protein: +++ | 2 |
  Urine Protein: ++++ | 1 |

9. Secondary Outcome: Doublet Cohort: Duration of Response (DOR)
Description: The DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) determined per RECIST v1.1 or death from any cause, whichever occurs first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 130 weeks
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered. Only responders (participants with CR or PR with confirmation of response by investigator) were analyzed in this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 7
months | 11.07 [3.647 to NA] — Upper limit of 95% confidence interval was not calculable due to insufficient number of participants with events at study closure.

10. Secondary Outcome: Doublet Cohort: Progression-Free Survival (PFS)
Description: The PFS is defined as the time from the first study drug administration to the date of the first documented disease progression or death due to any cause, whichever comes first.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 130 weeks
Population: All-treated population included all enrolled participants exposed to the study treatment, regardless of the amount of treatment administered.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 31
months | 5.95 [5.355 to 9.101]

11. Secondary Outcome: Doublet Cohort: Disease Control Rate (DCR)
Description: The DCR is defined as the percentage of participants who achieved confirmed CR, confirmed PR or stable disease (SD) as per RECIST v1.1. The SD is defined as neither sufficient shrinkage from the baseline study to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 130 weeks
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 31
percentage of participants | 83.9 [66.27 to 94.55]

12. Secondary Outcome: Triplet Cohort: Objective Response Rate
Description: The ORR is defined as percentage of participants with confirmed CR or PR as BOR determined per RECIST v1.1.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 130 weeks
Population: No participants were enrolled in the triplet cohort due to the early termination of the study.
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 0

13. Secondary Outcome: Doublet Cohort: Maximum Observed Concentration (Cmax) of Tusamitamab Ravtansine
Description: Blood samples were collected for the measurement of Cmax of tusamitamab ravtansine concentrations. Cmax of tusamitamab ravtansine was calculated using non-compartmental method.
Time Frame: Day 1 of Cycles 1 and 4
Population: The Pharmacokinetic (PK) population included all participants from the all-treated population with at least 1 post-baseline PK concentration with adequate documentation of dosing and sampling dates and times. Only participants analyzed and data collected at specific timepoints are reported.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 6
microgram per milliliter (mcg/mL)
  Cycle 1 Day 1 | 70.0 (11.9)
  Cycle 4 Day 1: number analyzed (Participants) | 4
  Cycle 4 Day 1 | 82.5 (16.3)

14. Secondary Outcome: Doublet Cohort: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 14 Days (AUC0-14d) of Tusamitamab Ravtansine
Description: Blood samples were collected for the measurement of AUC0-14d of tusamitamab ravtansine concentrations. AUC0-14d was calculated using the trapezoidal method from time 0 to 14 days and non-compartmental method.
Time Frame: Day 1 of Cycles 1 and 4
Population: The PK population included all participants from the all-treated population with at least 1 post-baseline PK concentration with adequate documentation of dosing and sampling dates and times. Only participants analyzed and data collected at specific timepoints are reported.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 6
day*mcg/mL
  Cycle 1 Day 1 | 312 (71.3)
  Cycle 4 Day 1: number analyzed (Participants) | 4
  Cycle 4 Day 1 | 459 (26.8)

15. Secondary Outcome: Doublet Cohort: Concentration Observed Before Treatment Administration During Repeated Dosing (Ctrough) of Ramucirumab
Description: Blood samples were collected for the measurement of Ctrough of ramucirumab concentrations. Ctrough was calculated using non-compartmental method.
Time Frame: Cycle 2 Day 1
Population: The PK population included all participants from the all-treated population with at least 1 post-baseline PK concentration with adequate documentation of dosing and sampling dates and times. Only participants analyzed and data collected at Cycle 2 Day 1 are reported.
Measure: Mean (Standard Deviation); unit: nanogram/mL
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 24
nanogram/mL | 32481.7 (11656.52)

16. Secondary Outcome: Number of Participants With Anti-Therapeutic Antibodies (ATAs) Against Tusamitamab Ravtansine
Description: Blood samples were collected to assess the presence of ATA against tusamitamab ravtansine in plasma from all participants. Treatment-emergent ATA is defined as participant with at least 1 treatment-induced/boosted ATA during the treatment period.
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Population: The ATA population included all participants from the all-treated population with at least 1 post-baseline ATA result (negative, positive, or inconclusive). No participants were enrolled in the triplet cohort due to the early termination of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 31 | 0
Participants | 4 |

17. Primary Outcome: Doublet Cohort - Part 1: Number of Participants With Study Drug-Related Dose-Limiting Toxicity (DLT)
Description: The following AEs occurred during the first 2 cycles of treatment, unless due to disease progression or to a cause obviously unrelated to study drug, were considered DLTs: • Grade 4 neutropenia for 7 or more consecutive days. • Grade 3 to 4 neutropenia complicated by fever. • Grade >=3 thrombocytopenia. • Elevated urine protein >=3 gram(g)/24 hour. • Grade 4 non-hematologic AE. • Grade >=3 keratopathy. • Grade 4 or refractory hypertension. In addition, any other AE that the Investigators and sponsor deemed to be dose limiting, regardless of its grade, was also considered as DLT.
Time Frame: From Cycle 1 Day 1 up to Cycle 2 Day 14, approximately 28 days
Population: DLT-evaluable (Part 1) population included all enrolled participants who received 2 cycles with at least 80% of the intended dose for both tusamitamab ravtansine and ramucirumab at each of the 2 first infusions unless they discontinued the study intervention before the end of Cycle 2 due to a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 6
Participants | 0

18. Primary Outcome: Doublet Cohort - Part 2: Objective Response Rate (ORR)
Description: The ORR is defined as percentage of participants with confirmed complete response (CR) or partial response (PR) as best overall response (BOR) determined per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. The CR is defined as disappearance of all target lesions. The PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumor assessments performed at baseline, and every 8 weeks +/-7 days thereafter, approximately 130 weeks
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab
Number analyzed (Participants) | 31
percentage of participants | 22.6 [9.59 to 41.10]

19. Primary Outcome: Triplet Cohort: Number of Participants With Study Drug-Related Dose-Limiting Toxicity
Description: The following AEs occurred during the first cycle of treatment, unless due to disease progression or to a cause obviously unrelated to study drug, were considered DLTs: • Grade 4 neutropenia for 7 or more consecutive days. • Grade 3 to 4 neutropenia complicated by fever. • Grade >=3 thrombocytopenia. • Elevated urine protein >=3 g/24 hour. • Grade 4 non-hematologic AE. • Grade >=3 keratopathy. • Grade 4 or refractory hypertension. In addition, any other AE that the Investigators and sponsor deemed dose limiting, regardless of its grade, was also considered as DLT.
Time Frame: From Cycle 1 Day 1 up to Cycle 1 Day 21
Population: No participants were enrolled in the triplet cohort due to the early termination of the study.
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug (Day 1) up to Day 30 post last dose of study drug, approximately 134 weeks
Description: Analysis was performed on all-treated population. No participants were enrolled in the triplet cohort due to the early termination of the study.
Groups:
- Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab: Participants were planned to receive tusamitamab ravtansine 150mg/m^2 plus ramucirumab 10 mg/kg and pembrolizumab 200 mgIV infusion every 3 weeks (Q3W) until disease progression, unacceptable AE, or the participant's or investigator's decision to stop the treatment.
Arm/Group | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 13/31 | 0/0
Serious Adverse Events (participants affected / at risk) | 7/31 | 0/0
Other Adverse Events (participants affected / at risk) | 31/31 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab (N=31) | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab (N=0)
Abscess Limb (Infections and infestations) | 1 (1) | NA
Pneumonia (Infections and infestations) | 1 (1) | NA
Cutaneous T-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | NA
Confusional State (Psychiatric disorders) | 1 (1) | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Colitis Ulcerative (Gastrointestinal disorders) | 1 (1) | NA
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | NA
Renal Impairment (Renal and urinary disorders) | 1 (1) | NA
Disease Progression (General disorders) | 1 (1) | NA
Multiple Organ Dysfunction Syndrome (General disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab (N=31) | Tusamitamab Ravtansine 100 mg/m^2 + Ramucirumab + Pembrolizumab (N=0)
Covid-19 (Infections and infestations) | 7 (7) | NA
Cystitis (Infections and infestations) | 3 (5) | NA
Rash Pustular (Infections and infestations) | 2 (2) | NA
Pyogenic Granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | NA
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | NA
Hypothyroidism (Endocrine disorders) | 2 (2) | NA
Decreased Appetite (Metabolism and nutrition disorders) | 9 (12) | NA
Delirium (Psychiatric disorders) | 2 (2) | NA
Dizziness (Nervous system disorders) | 3 (4) | NA
Dysgeusia (Nervous system disorders) | 5 (5) | NA
Headache (Nervous system disorders) | 7 (9) | NA
Neuropathy Peripheral (Nervous system disorders) | 4 (5) | NA
Paraesthesia (Nervous system disorders) | 4 (5) | NA
Cataract (Eye disorders) | 5 (6) | NA
Corneal Erosion (Eye disorders) | 2 (2) | NA
Dry Eye (Eye disorders) | 2 (2) | NA
Eye Pruritus (Eye disorders) | 2 (2) | NA
Keratitis (Eye disorders) | 2 (3) | NA
Keratopathy (Eye disorders) | 4 (7) | NA
Periorbital Oedema (Eye disorders) | 2 (2) | NA
Vision Blurred (Eye disorders) | 7 (11) | NA
Visual Acuity Reduced (Eye disorders) | 2 (2) | NA
Hypertension (Vascular disorders) | 10 (16) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (12) | NA
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | NA
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | NA
Constipation (Gastrointestinal disorders) | 6 (6) | NA
Diarrhoea (Gastrointestinal disorders) | 9 (9) | NA
Gingival Bleeding (Gastrointestinal disorders) | 3 (7) | NA
Nausea (Gastrointestinal disorders) | 13 (19) | NA
Vomiting (Gastrointestinal disorders) | 5 (7) | NA
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | NA
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (5) | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | NA
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | NA
Rash Pruritic (Skin and subcutaneous tissue disorders) | 3 (4) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | NA
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | NA
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | NA
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | NA
Proteinuria (Renal and urinary disorders) | 10 (19) | NA
Asthenia (General disorders) | 8 (12) | NA
Fatigue (General disorders) | 4 (4) | NA
Mucosal Inflammation (General disorders) | 3 (3) | NA
Oedema Peripheral (General disorders) | 5 (7) | NA
Pain (General disorders) | 2 (2) | NA
Pyrexia (General disorders) | 2 (2) | NA
Alanine Aminotransferase Increased (Investigations) | 3 (5) | NA
Aspartate Aminotransferase Increased (Investigations) | 3 (4) | NA
Gamma-Glutamyltransferase Increased (Investigations) | 2 (2) | NA
Neutrophil Count Decreased (Investigations) | 3 (23) | NA
Platelet Count Decreased (Investigations) | 7 (8) | NA

LIMITATIONS AND CAVEATS:
The study was prematurely terminated due to the discontinuation of the overall development of tusamitamab ravtansine (SAR408701) by the sponsor. The decision was not related to any safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT04394624/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04394624/SAP_001.pdf